CLINICAL TRIAL: NCT06557681
Title: The Effect of Virtual Reality Treadmill-Based Gait Training on Gait and Balance Ability in Chronic Stroke Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-2023-0088
Record Dates: First submitted 2024-08-08; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Stroke; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Receives conventional therapy (physical therapy)
  Interventions: Device: Virtual Reality-Treadmill Training Group (VTT)
- Control Group (Experimental): Receives conventional therapy (physical therapy)
  Interventions: Other: Conventional Therapy Group (CT)

INTERVENTIONS:
Device: Virtual Reality-Treadmill Training Group (VTT) — The Virtual Reality-Treadmill Training Group (VTT) will consist of 15 participants who will undergo 12 training sessions over 6 weeks, with each session occurring twice a week. Each session will include 30 minutes of conventional rehabilitation therapy followed by an additional 30 minutes of virtual reality-treadmill training. The sequence of these therapies can vary with each session. The virtual reality-treadmill training, conducted under the supervision of a therapist, will focus on five key components: precision stepping, obstacle negotiation, direction of progression, precision acceleration, and walking velocity. Evaluations of walking and balance abilities will be conducted before and after the intervention.
  Arms: Experimental Group
Other: Conventional Therapy Group (CT) — The Conventional Therapy Group (CT) will consist of 15 participants who will undergo 12 training sessions over 6 weeks, with each session occurring twice a week. Each session will include 30 minutes of conventional rehabilitation therapy, aimed at improving walking and balance functions. The therapy will be administered by a therapist and may include exercises focused on muscle strength increase, gait training for step length and walking speed improvement, and balance training. Evaluations of walking and balance abilities will be conducted before and after the intervention.
  Arms: Control Group

SUMMARY:
Walking independence is one of the most important goals for stroke patients and a major factor influencing their return to society after the onset of stroke. Stroke patients experience walking difficulties due to hemiplegia and have an increased risk of falls due to impaired balance ability. Recent studies have shown that treadmill-based walking training incorporating virtual reality can help improve walking and balance functions in actual stroke patients. However, there are few randomized clinical trials with control groups, highlighting the need for further research to ensure the reliability of clinical effects.

Therefore, this study aims to investigate the impact of treadmill-based training incorporating virtual reality on walking and balance functions. The training equipment to be used is the C-mill VR+ device, which enables walking training and assessment, balance training and assessment, and obstacle training using a front screen and treadmill videos. The investigators intend to thoroughly examine the walking ability and balance ability of the subjects obtained through this equipment, along with various evaluation tools.

ELIGIBILITY:
* Inclusion Criteria:

  1. Adult patients aged 19 years or older.
  2. Confirmed diagnosis of stroke by a neurologist or neurosurgeon through radiological methods such as CT or MRI.
  3. Chronic hemiplegic stroke patients, six months post-stroke onset.
  4. Patients with a Functional Ambulatory Category score of 3 or higher.
  5. Patients with a Mini-Mental State Examination (MMSE) score of 10 or higher, who understand the study, are willing to participate voluntarily, and have given consent to participate.
* Exclusion Criteria:

  1. Acute/subacute stroke patients within six months of stroke symptom onset.
  2. Patients with quadriplegia.
  3. Patients with ataxia.
  4. Patients with severe joint contracture of the lower limbs that makes wearing orthotics difficult.
  5. Patients with neurological, musculoskeletal, or cardiopulmonary diseases that affect walking.
  6. Any other cases deemed inappropriate for participation by the researcher.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-09-27 (Estimated); Study Completion 2024-09-27 (Estimated)

PRIMARY OUTCOMES:
Time Up and Go (TUG) | Pret-intervention Assessment
  The Timed Up and Go (TUG) test is a simple and reliable assessment used to evaluate a patient's mobility and balance abilities. During the test, the patient starts seated in a chair, then stands up, walks 3 meters to a designated marker, turns around, walks back to the chair, and sits down. The time taken to complete this sequence is measured. Shorter completion times indicate better mobility and balance. The TUG test is widely used to assess walking ability and fall risk in various conditions, including stroke and geriatric disorders.
Time Up and Go (TUG) | Baseline (Pre-intervention) and immediately after intervention completion (6 weeks after intervention start)
  The Timed Up and Go (TUG) test is a simple and reliable assessment used to evaluate a patient's mobility and balance abilities. During the test, the patient starts seated in a chair, then stands up, walks 3 meters to a designated marker, turns around, walks back to the chair, and sits down. The time taken to complete this sequence is measured. Shorter completion times indicate better mobility and balance. The TUG test is widely used to assess walking ability and fall risk in various conditions, including stroke and geriatric disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Department and Research Institute of Rehabilitation Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han SH, Jang HJ, Lee JW, Cheong JW, Kim YD, Nam HS, Kim DY. The effect of virtual reality-based treadmill gait training on functional mobility and balance in chronic stroke patients: a randomized controlled trial. Front Neurol. 2025 Jul 21;16:1603233. doi: 10.3389/fneur.2025.1603233. eCollection 2025. PMID 40761640